CLINICAL TRIAL: NCT06234930
Title: The Feasibility, Safety and Tolerability of Virtual Reality-based Audiovisual Stimulation
Brief Title: The Feasibility, Safety and Tolerability of VR-based Audiovisual Stimulation
Acronym: CFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clarity Health Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CHT0001
Record Dates: First submitted 2024-01-12; First posted 2024-01-31 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy Aging; Alzheimer's Disease
Keywords: Sensory neurostimulation; Non-invasive neuromodulation; Alzheimer's Disease; AD; Healthy; 50-90 years old; Gamma sensory stimulation; Virtual Reality; MCI
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Sham-controlled study where participants from two groups (Cognitively Impaired due to AD and Cognitively Healthy participants) are exposed to both active and sham conditions.
Who Masked: Participant
Masking Description: Participants will undergo sequential exposure to various stimulation conditions in a random order. The nature of each condition will not be disclosed to participants. The experimenter is unmasked to ensure protocol adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active and Sham Audiovisual Stimulation (Mild AD and MCI due to AD): (Experimental): Both active and sham stimulation conditions will be delivered to 25 cognitively impaired participants to demonstrate the mechanism of action of the intervention.
  Interventions: Device: Audiovisual stimulation VR system
- Active and Sham Audiovisual Stimulation (Cognitively Healthy): (Experimental): Both active and sham stimulation conditions will be delivered to 25 healthy participants to demonstrate the mechanism of action of the intervention.
  Interventions: Device: Audiovisual stimulation VR system

INTERVENTIONS:
Device: Audiovisual stimulation VR system — Delivery of synchronized auditory and visual stimuli at varying frequencies via a VR headset.
  Other Names: VR-based audiovisual stimulation; Sensory stimulation

SUMMARY:
This is a single-blind, sham-controlled, clinical trial that aims to evaluate the safety, tolerability, and feasibility of delivering audiovisual stimulation via a Virtual Reality (VR) headset to people cognitively impaired due to Alzheimer's and cognitively unimpaired people.

DETAILED DESCRIPTION:
Audiovisual stimulation is a non-invasive approach that uses synchronized light and sound stimuli to modulate neural activity and cognitive processes.

Recent literature suggests that when applied chronically, audiovisual stimulation may slow down the progression of Alzheimer's disease (AD). In contrast to traditional methods employing Light Emitting Diodes (LEDs) and computer screens for the delivery of visual stimuli, our study explores the feasibility, safety, and tolerability of delivering acute audiovisual stimulation via a Virtual Reality (VR) headset.

The investigators plan to recruit a total of 50 participants (n=25 mild AD or MCI due to AD and n=25 cognitively healthy participants). Audiovisual stimulation will be delivered over one experimental session to every participant. Stimuli will be embedded in passive environments and in a sound-video associative memory task. All participants will be exposed to stimulation at different frequencies and a sham condition will be used as a control. To determine the feasibility of VR-based audiovisual stimulation, the investigators will use electroencephalography (EEG) and measure the responsiveness of participants' brain activity to the acute intervention. Safety and tolerability will be evaluated using questionnaires.

This clinical trial aims to provide valuable insights into the development of a non-invasive therapy for early-stage Alzheimer's disease, while assessing the feasibility and safety of using VR technology to deliver audiovisual stimulation.

ELIGIBILITY:
Inclusion Criteria Mild AD/ MCI due to AD Participants:

* Age between 50 - 90 years old.
* A clinical diagnosis of Mild Cognitive Impairment due to Alzheimer's disease (confirmed by PET scan or CSF biomarkers) or Mild Alzheimer's disease
* MoCA score of 18-25.
* Willingness to sign informed consent document (if deemed to not have the capacity to sign the informed consent, a legally authorized representative will be asked to provide surrogate consent).
* Sufficient visual and hearing ability.
* Formal education of 8 or more years.
* Native English speakers or demonstrated fluency in English (participant; and LAR as needed)

Inclusion Criteria Cognitively Healthy Participants:

* Age between 50 - 90 years old.
* A MoCA score above or equal to 26.
* Willingness to sign informed consent document.
* Sufficient visual and hearing ability.
* Formal education of 8 or more years.
* Native English speakers or demonstrated fluency in English (participant)

Exclusion Criteria Mild AD/ MCI due to AD Participants:

* Previous exposure to monoclonal antibody medication (e.g., Lecanemab, Aducanumab).
* Active treatment with Memantine within the past 30 days.
* Initiation of acetylcholinesterase inhibitors within the past 30 days.
* A history of seizure or epilepsy including family history of seizure or epilepsy.
* A history of stroke.
* A diagnosis of migraine headache.
* History of alcohol use disorder within the past 2 years (DSM-V criteria).
* Current or past history of any neurological disorder other than dementia.
* Use of hearing aid device(s).
* Any known blood pathogens or disorders.
* Has any clinically significant medical disorder, condition, disease or clinically significant finding at screening that precludes participant's participation in study activities.
* Pregnancy (Verbal confirmation).
* Geriatric Depression Scale (GDS) >8

Exclusion Criteria Cognitively Healthy Participants:

* Active treatment with Memantine within the past 30 days.
* Initiation of treatment with acetylcholinesterase inhibitors (e.g., donepezil, rivastigmine and galantamine) within the past 30 days.
* A history of seizure or epilepsy including family history of seizure or epilepsy.
* A history of stroke.
* A diagnosis of migraine headache.
* History of alcohol use disorder within the past 2 years (DSM-V criteria).
* Use of hearing aid device(s).
* Any known blood pathogens or disorders.
* A diagnosis of Alzheimer's disease and related dementias.
* Has any clinically significant medical disorder, condition, disease or clinically significant finding at screening that precludes participant's participation in study activities.
* Pregnancy (Verbal confirmation)
* Geriatric Depression Scale (GDS) >8

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Changes in brain activity associated with exposure to VR-based audiovisual stimulation | Immediately after the intervention
  Feasibility of VR-based audiovisual stimulation will be assessed by quantifying significant changes in participants' brainwave activity during varying stimulation frequencies in comparison to baseline.
Level of tolerance to VR-based sensory stimulation exposure | Immediately after the intervention
  Tolerability will be assessed using a Likert scale ranging from 1 (indicating poor) to 7 (indicating good) to evaluate the overall VR-based sensory stimulation experience.
Incidence of Stimulation-Emergent Adverse Events | Immediately after the intervention
  Safety will be assessed via a questionnaire asking for any stimulation-related adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Reis, PhD, Principal Investigator — Clarity Health Technologies
Locations (2):
- United States (2):
  - The Sequoias Portola Valley, Portola Valley, California
  - Lakeview Institute of Clinical Research LLC, Leesburg, Florida

IPD SHARING:
Plan to Share IPD: No